CLINICAL TRIAL: NCT03323385
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, Evaluation of the Safety and Efficacy of Preoperative N1539 In Colorectal Surgery
Brief Title: Evaluation of Preoperative N1539 in Colorectal Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baudax Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REC-17-024
Record Dates: First submitted 2017-10-24; First posted 2017-10-27 (Actual); Results first posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-05

CONDITIONS: Pain, Postoperative
Keywords: Colorectal surgery; Pain; Analgesia; N1539; Phase 3b
MeSH Terms: conditions — Pain, Postoperative; Pain; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- N1539 30 mg (Experimental): N1539 (meloxicam injection for IV use) 30 mg every 24 hours
  Interventions: Drug: N1539
- IV Placebo (Placebo Comparator): IV Placebo every 24 hours
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N1539 — Once Daily
  Other Names: Intravenous meloxicam
  Arms: N1539 30 mg
Drug: Placebo — Once Daily
  Other Names: Intravenous placebo
  Arms: IV Placebo

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of preoperative dosing of N1539 30 mg in subjects undergoing colorectal surgery, including clinical laboratory tests, wound healing evaluation, incidence of anastomotic leaks, and incidence of Adverse Events (AEs) and Serious AEs (SAEs).

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily provide written informed consent.
* Be planned to undergo primary (no repeat procedures) open or laparoscopic colorectal surgery (laparoscopic expected to require a ≥ 5 cm incision) with bowel resection and/or anastomosis.
* ASA physical status category 1, 2, or 3.
* Female subjects not pregnant or planning/attempting to become pregnant, not lactating; or commits to the use of an acceptable form of birth control for the duration of the study.
* Have a body mass index <40 kg/m^2

Exclusion Criteria:

* Have a known allergy or hypersensitivity to any study treatment.
* Planned surgical procedure includes a resection beyond the peritoneal reflection, is related to an acute bout of diverticulitis, or is associated with an emergency procedure.
* Have a history of myocardial infarction within the preceding 12 months.
* Have, as determined by the investigator or the sponsor's medical monitor, a history or clinical manifestations of significant condition that would preclude participation.
* Have active or recent (within 6 months) gastrointestinal ulceration or bleeding, with exception of events related to an ulcerative colitis diagnosis.
* Have a known bleeding disorder which may be worsened with the administration of an NSAID.
* Be currently receiving treatment with oral meloxicam (Mobic®) or another NSAID within 48 hours prior to surgery.
* Have previously received N1539/IV meloxicam or received any investigational product within 30 days before dosing with study medication.
* Have undergone or be expected to undergo radiation therapy, chemotherapy, or other biological therapy for cancer treatment, within 60 days prior to screening through last follow-up.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2018-09-26 (Actual); Study Completion 2018-09-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Research Center, Florence, Alabama
  - Research Center, Mobile, Alabama
  - Research Center, Miami, Florida
  - Research Center, Tampa, Florida
  - Research Center, Metairie, Louisiana
  - Research Center, Jackson, Mississippi
  - Research Center, Cleveland, Ohio
  - Research Center, Columbus, Ohio
  - Research Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Silinsky JD, Marcet JE, Anupindi VR, Karkare SU, Shah DR, Mack RJ, McCallum SW, Du W, Freyer A, Black LK. Preoperative intravenous meloxicam for moderate-to-severe pain in the immediate post-operative period: a Phase IIIb randomized clinical trial in 55 patients undergoing primary open or laparoscopic colorectal surgery with bowel resection and/or anastomosis. Pain Manag. 2021 Jan;11(1):9-21. doi: 10.2217/pmt-2020-0061. Epub 2020 Oct 23. PMID 33094682

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | N1539 30 mg | IV Placebo
Started | 27 | 30
Dosed | 27 | 28
Completed | 26 | 27
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Noncompliance | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | N1539 30 mg | IV Placebo | Total
Number analyzed (Participants) | 27 | 28 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (11.18) | 60.6 (11.07) | 59.7 (11.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 15 | 17 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 22 | 23 | 45
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 27 | 28 | 55

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Safety and Tolerability - Number of Subjects With an AE
Description: Evaluate the incidence of adverse events in subjects receiving N1539 30 mg vs. placebo prior to colorectal surgery
Time Frame: Up to 30 days
Population: All randomized subjects
Measure: Number; unit: participants
Arm/Group | N1539 30 mg | IV Placebo
Number analyzed (Participants) | 27 | 28
participants | 23 | 26

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | N1539 30 mg | IV Placebo
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/28
Serious Adverse Events (participants affected / at risk) | 3/27 | 4/28
Other Adverse Events (participants affected / at risk) | 11/27 | 17/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N1539 30 mg (N=27) | IV Placebo (N=28)
Ileus (Gastrointestinal disorders) | 1 (1) | 2 (2)
Incision site cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Paranasal sinus benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N1539 30 mg (N=27) | IV Placebo (N=28)
Nausea (Gastrointestinal disorders) | 9 (11) | 14 (17)
Vomiting (Gastrointestinal disorders) | 5 (5) | 5 (5)
Ileus (Gastrointestinal disorders) | 1 (1) | 5 (5)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Urinary retention (Renal and urinary disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Discussion and/or publication of data generated is not permitted without the prior written consent of the sponsor.

DOCUMENTS (2):
  • Study Protocol (2017-11-16): https://cdn.clinicaltrials.gov/large-docs/85/NCT03323385/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-30): https://cdn.clinicaltrials.gov/large-docs/85/NCT03323385/SAP_001.pdf